CLINICAL TRIAL: NCT00514111
Title: Factors Associated to Success of Hepatitis C Therapy
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Alexandre Naime Barbosa, SAE e Hospital Dia de Aids - Faculdade de Medicina de Botucatu - Unesp
Other Study IDs: upeclin/HC/FMB-Unesp-16
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Hepatitis, Viral, Non-A, Non-B, Parenterally-Transmitted
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin; peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HVC Patients: HVC patients attended in SAE e HD.
  Interventions: Drug: pegylated-interferon, conventional-interferon, ribavirin

INTERVENTIONS:
Drug: pegylated-interferon, conventional-interferon, ribavirin — Genotype 1: pegylated-interferon 2a or 2b plus ribavirin for 48 weeks. Genotype 3: conventional-interferon 2a or 2b plus ribavirin for 24 weeks.
  Other Names: Pegasys; PegIntron; Ribavirin

SUMMARY:
The aim of this study is to evaluate the sustained virologic response (RVS) in HVC patients treated with pegylated-interferon or conventional-interferon and ribavirin, and to investigate the associated factors with RVS, by means of retrospective analysis.

DETAILED DESCRIPTION:
Chronic hepatitis C virus(HVC) is a major public-health problem since it presents a long phase of clinical latency which makes its early diagnosis difficult and results in the development of a large number of cases to complications such as cirrhosis, hepatic insufficiency and hepatocarcinoma. In Brazil, it is estimated three million estimated cases to 52 thousand reports. The aim of this study is to evaluate the sustained virologic response (RVS) in HVC patients treated with pegylated-interferon or conventional-interferon and ribavirin, and to investigate the associated factors with RVS, by means of retrospective analysis.

ELIGIBILITY:
Inclusion Criteria:

* HVC patients that received specific treatment with pegylated-interferon or conventional-interferon, and ribavirin

Exclusion Criteria:

* No HVC infection or treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HVC patients attended in SAE e HD.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre N Barbosa, MD, MSc, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- SAE e Hospital Dia de Aids, Botucatu, São Paulo, Brazil